CLINICAL TRIAL: NCT03816852
Title: Clinical Study on the Safety and Effectiveness of Human Umbilical Cord Mesenchymal Stem Cells in the Treatment of Premature Ovarian Insufficiency
Brief Title: The Safety and Efficiency Study of Mesenchymal Stem Cell (19#iSCLife®-POI) in Premature Ovarian Insufficiency
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Others
Sponsor: Sclnow Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCLnow-HNRM-01
Record Dates: First submitted 2019-01-17; First posted 2019-01-25 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Premature Ovarian Failure
Keywords: Premature Ovarian Failure; Premature Ovarian Insufficiency; mesenchymal stem cell
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dose group (Experimental): Intravenous infusion with hucMSCs, 9*10^7 cells, 30ml
  Interventions: Biological: hucMSCs
- Medium dose group (Experimental): Intravenous infusion with hucMSCs, 6*10^7 cells, 30ml
  Interventions: Biological: hucMSCs
- Low dose group (Experimental): Intravenous infusion with hucMSCs, 3*10^7 cells, 30ml
  Interventions: Biological: hucMSCs

INTERVENTIONS:
Biological: hucMSCs — Human umbilical cord mesenchymal stem cells were transplanted by intravenous infusion

SUMMARY:
Evaluate the safety of human umbilical cord mesenchymal stem cells (hucMSCs) in POI treatment; Evaluate the effective hucMSCs in POI treatment. Compare different infusion mode, meanwhile compare with hormone replacement therapy (HRT) withdrawal, so that assessing the stem cell therapy.

DETAILED DESCRIPTION:
Premature ovarian insufficiency (POI) or premature ovarian failure (POF), is the loss of function of the ovaries before age 40, which has the features of menstrual disorder with high gonadotropic hormone and low estrogen. The morbidity of POI is about 0.1% among woman before 40 years, 10-28% among woman with primary amenorrhea, and 4-18% among woman with secondary amenorrhea. Recent years research shows different sources of stem cell could be used to POI, and with effective results.

Above all, this experiment designed to as a single center, random, and control experiment. treat POI patients wit human umbilical cord mesenchymal stem cells (MSCs). After regular follow-up and analysis, assessing the safety and effective of MSCs in POI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic criteria of European Society of Human Reproduction and Embryology
* No hormonotherapy and chinese traditional medicine within 3 months;
* Understand and sign informed consent.

Exclusion Criteria:

* Patient with congenital adrenocortical hyperplasia;
* Patient with Cushing syndrome;
* Patient with Thyroid dysfunction;
* Patient with hyperprolactinemia;
* Patient with pituitary amenorrhea or hypothalamic amenorrhea;
* Patient with HIV, hepatitis;
* Gene defect (eg. Turner syndrome, fragile X syndrome)
* Serious drug allergy history;
* Suffering from thrombophlebitis, thromboembolism including venous thrombosis and arterial thrombosis;
* History of treatment of ovarian cysts or ovarian surgery
* With high tumor marker;
* Pregnant or lactating
* Receive other treatments that may affect the efficacy and safety of stem cells;
* Do not understand or without sign informed consent;
* The attending physician believes that it is not suitable for participating in this trial

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Menstrual changes | 270 days
  Observe the change of patients with irregular menstrual cycle

SECONDARY OUTCOMES:
Kupperman score | 270 days
  Mild: <14; moderate: 14-26; serious: >26
hormone level | 270 days
  Test the level change of Follicle-Stimulating Hormone (FSH), estrogen (E2), and Anti Mullerian Hormone (AMH)
Follicular development | 270 days
  Observe the size of ovarian follicles in each cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Guangzhi Liu, Dr, Study Director — Henan Provincial People's Hospital
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China